CLINICAL TRIAL: NCT00036764
Title: A Phase II Study Of Epothilone B Analog BMS 247550 (NSC # 710428) In Stage IV Malignant Melanoma
Brief Title: BMS-247550 in Treating Patients With Stage IV Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02464; NYU-0057; N01CM17103 (NIH); CDR0000069320 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2002-05-13; First posted 2003-01-27 (Estimated); Last update posted 2013-01-25 (Estimated); Status verified 2013-01

CONDITIONS: Recurrent Melanoma; Stage IV Melanoma
MeSH Terms: conditions — Melanoma | interventions — ixabepilone; Pharmacogenomic Testing

ARMS (1):
- Treatment (Experimental): Patients receive BMS-247550 IV over 1 hour on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: ixabepilone; Other: pharmacogenomic studies; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: ixabepilone — Given IV
  Other Names: BMS-247550; epothilone B lactam; Ixempra
Other: pharmacogenomic studies — Correlative studies
  Other Names: Pharmacogenomic Study
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Phase II trial to study the effectiveness of BMS-247550 in treating patients who have stage IV melanoma. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the efficacy of BMS-247550 in patients with stage IV melanoma. II. Determine the toxicity of this drug in these patients.

OUTLINE: This is a multicenter study. Patients are stratified according to the number of prior chemotherapy regimens (0 vs 1-2, including dacarbazine or temozolomide).

Patients receive BMS-247550 IV over 1 hour on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed stage IV melanoma
* At least 1 measurable lesion

  * Greater than 20 mm by conventional techniques
  * Greater than 10 mm by spiral CT scan
* Known brain metastases allowed if all of the following criteria are met:

  * Radiologically stable for at least 6 weeks after completion of whole brain radiotherapy
  * Stable at time of study
  * No mass effect present radiologically
  * No concurrent steroids to control symptoms of brain metastases
* Performance status - ECOG 0-2
* Performance status - Karnofsky 60-100%
* At least 3 months
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin normal
* AST/ALT no greater than 2.5 times upper limit of normal (ULN)
* Creatinine no greater than 1.5 times ULN
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No prior severe allergic reactions (grade III or IV or grade II not responsive to steroids) to taxanes or medications containing Cremophor EL
* No pre-existing grade 2 or greater peripheral neuropathy
* No HIV-positive patients receiving combination antiretroviral therapy
* No other concurrent uncontrolled illness
* No ongoing or active infection
* No psychiatric illness that would preclude study
* Prior vaccine therapy allowed
* Prior immunotherapy (e.g., interleukin-2 or interferon) allowed
* Stratum I:

  * No prior chemotherapy
* Stratum II:

  * No more than 2 prior chemotherapy regimens (must have included dacarbazine or temozolomide)
* See Disease Characteristics
* See Disease Characteristics
* Prior limb-perfusion therapy allowed (stratum II)
* No other concurrent investigational or commercial agents or therapies intended to treat malignancy
* No concurrent Hypericum perforatum

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2002-02; Primary Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
Response rate | Up to 2 years
  The 95% confidence intervals will be provided.

SECONDARY OUTCOMES:
Median time to progression | Time from the first day of treatment with BMS 247550 until the first documentation of disease progression, assessed up to 2 years
  Median time to progression will be described for each subgroup.
Incidence of related toxicities graded according to the revised NCI CTC version 2.0 | Up to 2 years
  Related toxicities will be described.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Pavlick, Principal Investigator — New York University Clinical Cancer Center
Locations (1):
- New York University Clinical Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Ott PA, Hamilton A, Jones A, Haas N, Shore T, Liddell S, Christos PJ, Doyle LA, Millward M, Muggia FM, Pavlick AC. A phase II trial of the epothilone B analog ixabepilone (BMS-247550) in patients with metastatic melanoma. PLoS One. 2010 Jan 20;5(1):e8714. doi: 10.1371/journal.pone.0008714. PMID 20098694